CLINICAL TRIAL: NCT03992807
Title: Patient-centered and Economic Effectiveness of a Decision Aid for Patients With Age-related Cataract: a Randomized Controlled Trial
Brief Title: A Decision Aid for Patients With Age-related Cataract
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019KYPJ090
Record Dates: First submitted 2019-06-11; First posted 2019-06-20 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Age-related Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A patient decision aid (Experimental): A patient decision aid that includes not only the standard general information, but also the quantitative risk information on the possible outcomes of cataract surgery as well as value clarification exercise.
  Interventions: Other: A patient decision aid
- A usual education booklet (Active Comparator): A traditional booklet with standard general information developed by the National Eye Institute (NEI) to help patients understand cataract.
  Interventions: Other: A usual education booklet

INTERVENTIONS:
Other: A patient decision aid — Potential participants receive a printed decision aid booklet with information about cataract surgery choice, and outcome data will be gathered using standardized questions in a structured interview after 2 weeks and 1 year.
  Arms: A patient decision aid
Other: A usual education booklet — Potential participants receive a usual booklet about cataract and cataract surgery, and outcome data will be gathered using standardized questions in a structured interview after 2 weeks and 1 year.
  Arms: A usual education booklet

SUMMARY:
To determine whether a decision aid increases informed decision about cataract surgery for patients with age-related cataract.

DETAILED DESCRIPTION:
The need for cataract surgery is on the rise globally due to the aging population and high demands for greater visual functioning. Patients with age-related cataract face their initial decision about when to undergo cataract surgery. Although the majority of patients want to participate in a shared decision-making process, no decision aid has been available to improve the quality of decision. The purpose of this study is to determine whether a decision aid increases informed decision about cataract surgery for patients with age-related cataract.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 50-80 years who have been resident in the selected study district for more than six months;
2. A definite diagnosis of age-related cataract;
3. Having not received cataract surgery;
4. Willing to participate in the study and provide informed content.

Exclusion criteria

1. Bilateral blindness (presenting distance visual acuity worse than 3/60);
2. Having ocular, hearing or mental disorder precluding reading or telephone interview;
3. Ocular disorders other than cataract leading to permanent vision loss that could not be corrected through cataract surgery;
4. Having cataract surgery contraindication.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2020-11-12 (Estimated)

PRIMARY OUTCOMES:
Informed choice about cataract surgery (the proportion of participants who make an informed choice，which is defined as a good knowledge score and an intention that is consistent with their attitude score) | 2 weeks post intervention
  Informed choice is an aggregated measure of multiple measurements, including knowledge (a 12-item questionnaire that assesses conceptual (items 1-10) and numerical (items 11-12) knowledge), attitudes (6 items, with 5 responses for each), and intentions (single item with 5 responses)
  Analysis: Informed Choice= Good Knowledge (score ≥50% in basic knowledge, ≥40% in knowledge associated with each treatment option, and at least 1 point in each numerical knowledge question) AND Positive Attitude (score ≥24) AND Positive Intention ("definitely will" or "likely to"), OR Good Knowledge AND Negative Attitude (score <23) AND Negative Intention ("unsure", "not likely to", or "definitely will not")

SECONDARY OUTCOMES:
Perceived importance of surgical benefit/harms | 2 weeks post intervention
  Purpose-developed items will be used to ask participants about their personal perceptions of the importance of specific outcomes in their decision-making about cataract surgery.
Perceived personal chances of surgical benefit/harms | 2 weeks post intervention
  Participants will be asked about their perceived personal likelihood of experiencing specific outcomes if they have cataract surgeries, compared with an average patient who had undergone cataract surgery.
Decisional conflict | 2 weeks post intervention
  Decisional conflict will be assessed using a 16-item Decisional Conflict Scale.
Decisional confidence | 2 weeks post intervention
  Decisional confidence will be assessed using a 11-item Decision Self Efficacy Scale.
Time perspective | 2 weeks post intervention
  This will be assessed using a 4-item short form of the Consideration of Future Consequences Scale, with five response categories ranging from strongly agree to strongly disagree.
Anticipated regret | 2 weeks post intervention
  Two items from a validated scale will measure anticipated regret about having cataract surgery (action regret) and about not having cataract (inaction regret).
Cataract worry and anxiety | 2 weeks post intervention
  A validated single item will measure participants' level of worry about progression of cataract, using four verbal response categories ranging from not worried at all to very worried. Anxiety will be measured with a six-item short form.
Booklet utilization and acceptability | 2 weeks post intervention
  Acceptability and utilization of materials will be assessed based on the following items:
  1. the proportion of participants who could read the booklet all the way through;
  2. the proportion of participants who agree that the information is new;
  3. the proportion of participants who agree that the length is just about right;
  4. the proportion of participants who think the information is balanced;
  5. the proportion of participants who agree that the booklet is clear and easy to understand;
  6. the proportion of participants who find the materials helpful;
  7. the proportion of participants who feel it worth recommending to others.
Undergoing cataract surgery | 1 year post intervention
  Self-reported undergoing cataract surgery will be assessed via telephone survey at 1 year.
Decision regret | 1 year post intervention
  The Decision Regret Scale will measure participants' level of regret regarding their initial decision whether to have cataract surgery or not.
Visual functioning | Baseline, 1 year post intervention
  This will be assessed using the Catquest 9SF questionnaire.
Fall questionnaire | 1 year post intervention
  This will be assessed using a single item question "Did you have any fall in the past 12 months whereby you landed on the ground or floor?"
Heath-related quality of life: Chinese version of the EQ-5D-5L telephone interview script | Baseline, 1 year post intervention
  This will be assessed using the simplified Chinese version of the EQ-5D-5L telephone interview script from the EuroQol research foundation.
Costs | Baseline, 1 year post intervention
  This will be assessed using the Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Flaxman SR, Bourne RRA, Resnikoff S, Ackland P, Braithwaite T, Cicinelli MV, Das A, Jonas JB, Keeffe J, Kempen JH, Leasher J, Limburg H, Naidoo K, Pesudovs K, Silvester A, Stevens GA, Tahhan N, Wong TY, Taylor HR; Vision Loss Expert Group of the Global Burden of Disease Study. Global causes of blindness and distance vision impairment 1990-2020: a systematic review and meta-analysis. Lancet Glob Health. 2017 Dec;5(12):e1221-e1234. doi: 10.1016/S2214-109X(17)30393-5. Epub 2017 Oct 11. PMID 29032195
- [Background] Kessel L, Andresen J, Erngaard D, Flesner P, Tendal B, Hjortdal J. Indication for cataract surgery. Do we have evidence of who will benefit from surgery? A systematic review and meta-analysis. Acta Ophthalmol. 2016 Feb;94(1):10-20. doi: 10.1111/aos.12758. Epub 2015 Jun 3. PMID 26036605
- [Background] McCarty CA, Keeffe JE, Taylor HR. The need for cataract surgery: projections based on lens opacity, visual acuity, and personal concern. Br J Ophthalmol. 1999 Jan;83(1):62-5. doi: 10.1136/bjo.83.1.62. PMID 10209437
- [Derived] Zheng Y, Qu B, Jin L, Wang C, Zhong Y, He M, Liu Y. Patient-centred and economic effectiveness of a decision aid for patients with age-related cataract in China: study protocol of a randomised controlled trial. BMJ Open. 2020 May 18;10(5):e032242. doi: 10.1136/bmjopen-2019-032242. PMID 32430445